CLINICAL TRIAL: NCT02707146
Title: Aligning the Visit Priorities of Complex Patients and Their Primary Care Providers
Brief Title: Aligning Patients and Their Primary Care Providers
Acronym: APP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CN-14-2070-H
Record Dates: First submitted 2016-03-04; First posted 2016-03-14 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Primary Health Care; Quality of Health Care; Comorbidity; Communication; Medical Informatics Applications
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tablet in the waiting room (Experimental): Patients in the intervention arm will be met in the waiting room prior to their primary care visit and will use the "Visit Planner" tool application on the tablet
  Interventions: Behavioral: Visit Planner; Device: iPad
- Health Education Handout (Active Comparator): Patients in the control arm will be met in the waiting room prior to their primary care visit and will be given an educational pamphlet on health lifestyle to review
  Interventions: Other: Attention Control Pamphlet

INTERVENTIONS:
Behavioral: Visit Planner — The Visit Planner is an application hosted on an iPad that guides the patient in preparing for the primary care visit
  Arms: Tablet in the waiting room
Other: Attention Control Pamphlet — Patients in the attention control arm will receive an approved educational handout on health lifestyle
  Arms: Health Education Handout
Device: iPad
  Arms: Tablet in the waiting room

SUMMARY:
This project focuses on improving the patient-provider primary care visit interaction by addressing the need to align patient and provider priorities in a way that incorporates patients' goals and preferences while supporting the clinical work of their providers.

DETAILED DESCRIPTION:
The aim of this clinical trial is to enroll new and/or complex patients and their physicians in a 12-month randomized study. At each scheduled primary care visit during the trial period, Intervention Patients will be provided with a waiting room Tablet loaded with the "Visit Planner" intervention tool designed to support prioritization and discussion of top health care concerns. Control Patients will be given a written educational handout to review. Patient-centered outcomes will be obtained at baseline and after visits using validated survey instruments. Clinical outcomes focus on differences in quality of care. If successful, this approach to aligning patient and provider visit priorities can potentially be disseminated and adapted to a wide variety of different care settings.

ELIGIBILITY:
Inclusion Criteria:

* Kaiser Permanente member with an assigned primary care provider, with at least one quality care gap at baseline (overdue screening tests, elevated risk factor levels, sub-optimal adherence to chronically prescribed medicines, current smoker)
* Patients must be either:

  * 1) relatively new to their provider (0-3 visits in past 18 months) or if associated with their provider for > 18 months,
  * 2) have evidence for medical complexity (4 or more prescribed medicines, in a chronic disease management program, or recently admitted to hospital or emergency department)

Exclusion Criteria:

* Excluded by their primary care provider

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2016-03; Primary Completion 2017-07 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Grant, MD MPH, Principal Investigator — Division of Research, KPNC
Locations (1):
- Oakland Medical Center, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grant RW, Lyles C, Uratsu CS, Vo MT, Bayliss EA, Heisler M. Visit Planning Using a Waiting Room Health IT Tool: The Aligning Patients and Providers Randomized Controlled Trial. Ann Fam Med. 2019 Mar;17(2):141-149. doi: 10.1370/afm.2352. PMID 30858257
- [Result] Kowalski CP, McQuillan DB, Chawla N, Lyles C, Altschuler A, Uratsu CS, Bayliss EA, Heisler M, Grant RW. 'The Hand on the Doorknob': Visit Agenda Setting by Complex Patients and Their Primary Care Physicians. J Am Board Fam Med. 2018 Jan-Feb;31(1):29-37. doi: 10.3122/jabfm.2018.01.170167. PMID 29330237
- [Result] Lyles CR, Altschuler A, Chawla N, Kowalski C, McQuillan D, Bayliss E, Heisler M, Grant RW. User-Centered Design of a Tablet Waiting Room Tool for Complex Patients to Prioritize Discussion Topics for Primary Care Visits. JMIR Mhealth Uhealth. 2016 Sep 14;4(3):e108. doi: 10.2196/mhealth.6187. PMID 27627965
- [Result] Ruvalcaba D, Nagao Peck H, Lyles C, Uratsu CS, Escobar PR, Grant RW. Translating/Creating a Culturally Responsive Spanish-Language Mobile App for Visit Preparation: Case Study of "Trans-Creation". JMIR Mhealth Uhealth. 2019 Apr 5;7(4):e12457. doi: 10.2196/12457. PMID 30950803
- [Derived] Santo EC, Vo MT, Uratsu CS, Grant RW. Patient-Defined Visit Priorities in Primary Care: Psychosocial Versus Medically-Related Concerns. J Am Board Fam Med. 2019 Jul-Aug;32(4):513-520. doi: 10.3122/jabfm.2019.04.180380. PMID 31300571

RESULTS

PARTICIPANT FLOW:
Groups:
- Tablet in the Waiting Room: Patients in the intervention arm will be met in the waiting room prior to their primary care visit and will use the "Visit Planner" tool application on the tablet
  Visit Planner: The Visit Planner is an application hosted on an iPad that guides the patient in preparing for the primary care visit
  iPad
Period: Overall Study
Arm/Group | Tablet in the Waiting Room | Health Education Handout
Started | 359 | 391
Completed | 359 | 388
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tablet in the Waiting Room | Health Education Handout | Total
Number analyzed (Participants) | 359 | 391 | 750
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 195 | 212 | 407
  >=65 years | 164 | 179 | 343
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (12.1) | 61.2 (11.7) | 60.8 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 235 | 251 | 486
  Male | 124 | 140 | 264
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: African-American | 115 | 97 | 212
  Race/ethnicity: Asian | 20 | 34 | 54
  Race/ethnicity: Hispanic | 69 | 98 | 167
  Race/ethnicity: Other (>1 race/ethnicity) | 14 | 15 | 29
  Race/ethnicity: White | 141 | 147 | 288
Region of Enrollment [Number; unit: participants]
  United States | 359 | 391 | 750

OUTCOME MEASURES:

1. Primary Outcome: Aggregate Measure of Guideline-Based Clinical Care Gaps
Description: All patients enrolled in the study will have one or more guideline-based care gaps at baseline. Care gaps are defined as: overdue for cancer screening (mammography, colorectal cancer), overdue for chronic disease monitoring (blood pressure, HbA1c), above goal for chronic disease (SBP > 140, HbA1c > 8%), or medication related (not prescribed a statin if clinically indicated, not prescribed medicine for osteoporosis if indicated, < 80% adherence to medication for diabetes, hypertension, or hyperlipidemia), or current smoker. The investigators will assess % of patients resolving baseline clinical care gaps after 12 months. The aggregate outcome will be defined as yes/no resolution of baseline care gap. The study arms will be compared using an aggregate measure of these guideline-based clinical care gaps.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tablet in the Waiting Room | Health Education Handout
Number analyzed (Participants) | 359 | 388
Participants | 184 | 210

2. Secondary Outcome: Patient-reported Outcomes
Description: Telephone survey will be conducted within 1 week of visit using validated questionnaire items that assess patient-provider communication and patient satisfaction with care
Time Frame: Within 1 week of primary care study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Tablet in the Waiting Room | Health Education Handout
Number analyzed (Participants) | 333 | 357
Participants
  Prepare list of questions? | 198 | 160
  Tell your doctor your top concerns at beginning o | 304 | 297
Statistical Analysis 1: Comparison: Tablet in the Waiting Room vs Health Education Handout; Test type: Superiority; Chi-squared; Odds Ratio (OR) = 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Tablet in the Waiting Room | Health Education Handout
All-Cause Mortality (participants affected / at risk) | 0/359 | 0/391
Serious Adverse Events (participants affected / at risk) | 0/359 | 0/391
Other Adverse Events (participants affected / at risk) | 0/359 | 0/391

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT02707146/Prot_SAP_000.pdf